CLINICAL TRIAL: NCT02505984
Title: Testing the Efficacy of Intranasal Oxytocin for the Prevention of Postpartum Depression and PTSD
Brief Title: Preventing Postpartum Depression With Intranasal Oxytocin
Acronym: IN-OXT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sharon Dekel, PhD, Assistant Professor in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2015P001100; 224421 (Other Grant/Funding Number: Claflin Distinguished Scholar Award); 225686 (Other Grant/Funding Number: Brain & Behavior Research Foundation); 1R21HD090396-01A1 (NIH)
Record Dates: First submitted 2015-07-19; First posted 2015-07-22 (Estimated); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Depression, Postpartum; Anxiety
Keywords: oxytocin, bonding; child development
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Active Comparator): Sub-group of participants receiving oxytocin nasal spray (Syntocinon)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Sub-group of participants receiving placebo nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Study participants will be randomized to a placebo or drug group.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — Study participants will be randomized to a placebo or drug group.
  Other Names: Salt solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to test a new treatment for preventing childbirth-related mental illness in postpartum mothers. The treatment is aimed at enhancing maternal bonding, reducing postpartum depression (PPD) and anxiety in mothers at risk, and promoting child development. To this end, the investigators will test the clinical utility of intranasal (IN) oxytocin (OXT) administered to mothers during the first postpartum days.

DETAILED DESCRIPTION:
Postpartum depression (PPD) is a debilitating disorder which imposes a threat to mother and infant health. An estimated 600,000 American women suffer from PPD annually, making it one of the most frequent complications of pregnancy. Available secondary preventive interventions are often ineffective, which calls for identifying novel means for prevention. Impaired mother-infant bonding is a hallmark of PPD. Depressed mothers may have difficulties developing maternal feelings and providing sensitive care. In turn, impaired bonding may worsen mother's depression. Conventional pharmacotherapy does not help with bonding impairment.

This study will attempt to fill in the current gap in effective preventive interventions for pregnant mothers at risk. Evidence in postpartum mothers indicates that high peripartum OXT levels are associated with enhanced maternal behavior and low levels with depression. Data also indicates that in depressed mothers, OXT levels may decrease during the first days following childbirth rather than increase as is the norm. Therefore, the investigators will test the therapeutic effects of OXT in women at risk for PPD. It is hypothesized that administration of IN-OXT (total daily dose 48 IU) over the course of four days from as early as day one postpartum in comparison to placebo will 1) enhance mother-infant bonding, 2) reduce depressive and anxiety symptoms at 5 days postpartum, and 3) facilitate child development.

ELIGIBILITY:
Inclusion Criteria:

* Third-trimester pregnant women being followed at the Massachusetts General Hospital (MGH) Obstetrics Program
* At risk of postpartum depression (PPD)

Exclusion Criteria:

* Failure to participate in regular prenatal check-ups
* Current diagnosis Diagnostic and Statistical Manual of Mental Disorders (DSM-5) mental disorder pertaining to psychosis or substance abuse
* Suicidality
* Obstetric complication (e.g., preeclampsia, excessive hemorrhaging)
* Use of potentially confounding or interacting medications
* Complicating pediatric medical condition in the newborn

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Dekel, PhD, Principal Investigator — Massachusetts General Hosptial
Locations (1):
- Massachusetts General Hosptial, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mah BL, Bakermans-Kranenburg MJ, Van IJzendoorn MH, Smith R. Oxytocin promotes protective behavior in depressed mothers: a pilot study with the enthusiastic stranger paradigm. Depress Anxiety. 2015 Feb;32(2):76-81. doi: 10.1002/da.22245. Epub 2014 Feb 12. PMID 24523054
- [Background] Skrundz M, Bolten M, Nast I, Hellhammer DH, Meinlschmidt G. Plasma oxytocin concentration during pregnancy is associated with development of postpartum depression. Neuropsychopharmacology. 2011 Aug;36(9):1886-93. doi: 10.1038/npp.2011.74. Epub 2011 May 11. PMID 21562482
- [Background] Fewtrell MS, Loh KL, Blake A, Ridout DA, Hawdon J. Randomised, double blind trial of oxytocin nasal spray in mothers expressing breast milk for preterm infants. Arch Dis Child Fetal Neonatal Ed. 2006 May;91(3):F169-74. doi: 10.1136/adc.2005.081265. Epub 2005 Oct 13. PMID 16223754
- [Background] Riem MM, Bakermans-Kranenburg MJ, Pieper S, Tops M, Boksem MA, Vermeiren RR, van Ijzendoorn MH, Rombouts SA. Oxytocin modulates amygdala, insula, and inferior frontal gyrus responses to infant crying: a randomized controlled trial. Biol Psychiatry. 2011 Aug 1;70(3):291-7. doi: 10.1016/j.biopsych.2011.02.006. Epub 2011 Apr 5. PMID 21470595
- [Background] Jobst A, Krause D, Maiwald C, Hartl K, Myint AM, Kastner R, Obermeier M, Padberg F, Brucklmeier B, Weidinger E, Kieper S, Schwarz M, Zill P, Muller N. Oxytocin course over pregnancy and postpartum period and the association with postpartum depressive symptoms. Arch Womens Ment Health. 2016 Aug;19(4):571-9. doi: 10.1007/s00737-016-0644-2. Epub 2016 Jun 20. PMID 27320943
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Massachusetts General Hospital Outpatient Obstetrics Clinic between January 2016 and December 2019. The first participant was enrolled on January 8, 2016, and the last participant was enrolled on December 4, 2019.
Pre-assignment Details: Of 56 enrolled participants, 42 were randomized to treatment.
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 20 | 22
Completed | 18 | 20
Not Completed | 2 | 2
Not completed — Enrolled in study under IRB Other Event (depression screening score below inclusion criteria) | 1 | 0
Not completed — Unreliable self-report data | 1 | 0
Not completed — Study blind opened during assessment | 0 | 1
Not completed — Noncompliance with study protocol | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.75 (5.27) | 32.59 (6.11) | 31.71 (5.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Non-Hispanic White | 14 | 11 | 25
  Black or African American | 3 | 2 | 5
  Asian or Asian American | 1 | 4 | 5
  Unknown | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
Screening Edinburgh Postnatal Depression Scale Score [Mean (Standard Deviation); unit: score on a scale] — Self-reported assessment of severity of maternal depression symptoms (higher scores mean worse outcome, range 0 - 30).
  score on a scale | 13.25 (3.73) | 13.23 (3.44) | 13.24 (3.53)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Effect on Mother-infant Bonding
Description: Day 5 postpartum:
  Self-report assessment of maternal bonding (Maternal Attachment Inventory, higher scores means better outcome, range 26 -104)
  2 months postpartum: Quantitative observational assessment of mother-infant bonding (Coding Interactive Behavior; mean score represents mean score of the study sample. Negative bonding includes age-appropriate items on maternal intrusiveness, infant withdrawal, and dyad negative sub-scales, higher scores indicate higher levels of negative bonding behavior (deviation above the mean represent worse outcome); positive bonding includes maternal sensitivity, maternal limit setting, infant involvement, and dyad reciprocity sub-scales, higher scores indicate higher levels of bonding behavior, deviation above the mean represent better outcome); and repeat of self-report (MAI)
Time Frame: 5 days and 2 months postpartum (on average)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
score on a scale
  Maternal bonding, 5 days postpartum | 99.33 (6.15) | 99.35 (6.92)
  Maternal bonding, 2 months postpartum | 101.11 (5.58) | 97.90 (7.28)
  Mother-infant bonding, 2 months postpartum (Observed, negative bonding, Z score) | -0.22 (0.81) | 0.20 (0.50)
  Mother-infant bonding, 2 months postpartum (Observed, positive bonding, Z score) | 0.19 (0.82) | -0.17 (0.59)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.093, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.077, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Treatment Effect on Maternal Depression Symptoms
Description: Self-reported assessment of severity of maternal depression symptoms (Edinburgh Postnatal Depression Scale, higher scores mean worse outcome, range 0 - 30).
Time Frame: Baseline and 5 days postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
score on a scale
  Maternal depression, pregnancy | 13.22 (2.98) | 13.35 (3.53)
  Maternal depression, 5 days postpartum | 7.72 (5.12) | 9.45 (5.49)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority; p > 0.9, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Treatment Effect on Maternal Anxiety Symptoms
Description: Self-reported severity of maternal anxiety symptoms (Brief Symptom Inventory, Anxiety sub-scale, higher scores means worse outcome, range 0 - 24).
Time Frame: Baseline and 5 days postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
score on a scale
  Maternal anxiety, pregnancy | 5.67 (5.55) | 6.95 (5.77)
  Maternal anxiety, 5 days postpartum | 5.44 (6.71) | 6.30 (6.74)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.8, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Child Development
Description: Quantitative observational assessment of infant communication, cognitive, and motor development (Bayley Scales of Infant Development, screening, higher scores better outcome, ranges for each subscale are reported for infants 1-6 months old (items are scored either 0 or 1) - communication scale range 0-4, cognitive scale range 0-7, motor scale range 0-12; note: Bayley Scales can be performed for up to 42 months old infants; developmentally advanced infants may achieve scores above the reported range scale above)
Time Frame: 2 months postpartum (on average)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 18 | 20
score on a scale
  Infant communication subscale, 2 months postpartum | 3.44 (0.78) | 3.55 (0.69)
  Infant cognition subscale, 2 months postpartum | 5.19 (1.21) | 5.61 (1.30)
  Infant motor subscale, 2 months postpartum | 6.88 (3.24) | 7.73 (3.11)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.7, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 14 weeks (on average)
Description: Study drug diary asked participants to report and list symptoms experienced, if applicable.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 3/20 | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=20) | Placebo (N=22)
Uterine Cramping (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Slight nosebleeding (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Chest tightness (Cardiac disorders) | 0 (0) | 1 (1) — Participant reported tightness in chest (unknown effect) after 1 dose; she was unsure if related to nasal spray. Event reported to Institutional Review Board (expedited review). Study blind was opened and identified participant as randomized placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT02505984/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT02505984/SAP_001.pdf
  • Informed Consent Form (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT02505984/ICF_002.pdf